CLINICAL TRIAL: NCT07287800
Title: A Prospective Study of Testosterone Supplementation in Hypogonadal Patients Receiving a Renal Transplant
Brief Title: TRT as an Adjunctive ERAS Therapy in ESRD Patients Undergoing Kidney Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nima Nassiri, Assistant Clinical Professor of Urology, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-5575; PATS 20252050 (Other Grant/Funding Number: American Urologic Association)
Record Dates: First submitted 2025-12-01; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hypogonadism, Male; End Stage Renal Disease (ESRD); Kidney Transplant
Keywords: ESRD; testosterone replacement therapy; hypogonadal; kidney transplant
MeSH Terms: conditions — Eunuchism; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone Replacement Therapy (Experimental)
  Interventions: Drug: Testosterone Replacement Therapy
- No Testosterone Replacement Therapy (No Intervention)

INTERVENTIONS:
Drug: Testosterone Replacement Therapy — Testosterone Replacement Therapy
  Arms: Testosterone Replacement Therapy

SUMMARY:
This prospective study aims to evaluate the safety and efficacy of testosterone replacement therapy (TRT) as an adjunct to an enhanced recover after surgery (ERAS) protocol in men with end-stage renal disease (ESRD) undergoing kidney transplantation.

Participants will be highly-listed hypogonadal men, defined as total testosterone level <300 on two occasions with clinical symptoms of hypogonadism, with ESRD who are expected to receive a kidney transplant within 6 months. Participants will be started on TRT, ideally for at least 3 months prior transplantation. The investigators will perform a subset analysis to evaluate if there is a significant difference in our endpoints by comparing these two subgroups (Three months or more receiving TRT vs. Less than three months receiving TRT). There will be no cut-off time for pre-transplant TRT. Following the intervention period, a historical control cohort of age-matched and health-matched patients will be identified, who have followed a standard transplant protocol that does not incorporate TRT. The primary outcome will evaluate safety, including 30- and 90-day adverse events, 3, 6, and 12-month allograft survival, and overall patient survival. Secondary outcomes will focus on (1) qualitative assessments of symptoms using validated questionnaires, (2) quantitative improvements in the hormonal profile before and after initiation of TRT and surgery, and (3) allograft function and incidence of delayed graft function. The results of this study could provide novel insights into the benefits of TRT in improving surgical outcomes in men with ESRD undergoing kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male patients older than 18 years old with confirmed end-stage renal disease (ESRD).
* Hypogonadal (testosterone level <300 ng/dL) with clinical symptoms of hypogonadism.
* Expected to undergo kidney transplantation within a 6-month period.
* Able and willing to comply with study procedures and follow-up visits.

Exclusion Criteria:

* Women or non-hypogonadal men.
* Any contraindications to testosterone therapy, including:

  * History of Breast Cancer
  * Severe untreated OSA
  * Polycythemia (Hct >54%)
  * Uncontrolled chronic heart failure (CHF)
  * A history of a Major Adverse Cardiac Event (MACE) within the past 6 months
  * Interest in fertility within 1 year
  * An unevaluated PSA >4.0 ng/mL or a PSA >3.0 ng/mL in individuals with risk factors for prostate cancer defined as:

    * Men with African ancestry
    * Men with first-degree relative with prostate cancer
    * Known genetic mutations including BRCA1/2
    * A history of Lynch Syndrome
    * Abnormal DRE
* Participants already receiving testosterone or other androgen therapies.
* Severe cardiovascular or pulmonary conditions that pose a high surgical risk.
* Any condition that, in the opinion of the investigator, would make the subject ineligible for the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 18 months
  Complications categorized by the CTCAE classification (grades 1-5)
Overall Survival | 18 months
  measured as a rate
Death-Censored- Graft Survival | 18 months
  Graft Survival will be the duration from transplantation until graft failure. Graft failure defined as (1) resumption of dialysis (2) allograft removal or (3) need for retransplantation/relisted on the transplant list
Healthcare Utilization Metrics | 18 months
  Hospital readmission rates
Length of hospitalization | 18 months
  days

SECONDARY OUTCOMES:
Serum Creatinine Levels | At 3-, 6-, and 12-months post-transplantation
  measured as mg/dL
estimated glomerular filtration rate (eGFR) | At 3-, 6-, and 12-months post-transplantation
  ml/min/1.73 m^2
Rate of delayed graft function | 1 week following transplant
  Defined as the need for dialysis within the first week post-transplant.
Tacrolimus trough level | 1 month after TRT initiation, and at 3-, 6-, and 12-months post-transplant
  ng/mL
Follicle-Stimulating Hormone (FSH) | Once prior to initiation of TRT surgery
  mIU/mL
Serum Testosterone Panel | Every 3 months after starting TRT; at the time of transplantation; 30-, 90-, 180-, 270-, and 360-days post transplantation
  Total, Free, and Bioavailable Testosterone Levels, measured as ng/dL
Prostate Specific Antigen (PSA) | at baseline prior to TRT therapy, and every 3-6 months during active hormone therapy.
  ng/mL
Luteinizing Hormone (LH) | Once prior to initiation of TRT surgery
  mIU/mL
Prolactin | Once prior to initiation of TRT surgery
  ng/mL
Hemoglobin | 1 month after TRT initiation, and at 3-, 6-, and 12-month intervals
  To assess for polycythemia, measured as g/dL
Hematocrit | 1 month after TRT initiation, and at 3-, 6-, and 12-month intervals
  To assess for polycythemia, measured as L/L, read as a percentage
Muscle Body Composition Analysis | at time of consent, 30 days, 180-days, and 360 days after transplantation
  SECA Body Analysis is a non-invasive scan measuring BMI, Fat-Mass Index, Fat Mass Percentage, Skeletal Muscle Mass, and Skeletal Muscle Mass Percentage
Qualitative Assessment of Hypogonadal Symptoms | at time of consent; every 3-6 months starting TRT; 30- and 90-days following transplantation
  qADAM is a validated questionnaire of 10 questions to assess hypogonadal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT07287800/Prot_SAP_000.pdf